CLINICAL TRIAL: NCT06450236
Title: An Open-label, Balanced, Randomized, Two Treatment, Two Sequence, Two Period, Two Way Cross-over, Single Dose Bioequivalence Study of Perampanel Tablets 10 mg of Humanis Sağlık A.Ş., Turkey and Fycompa 10 mg Film-coated Tablets of Eisai GmbH Edmund-Rumpler-Straße 3 60549 Frankfurt am Main Deutschland in Normal, Healthy, Adult, Human Subjects Under Fasting Condition
Brief Title: Bioequivalence Study of Perampanel Tablets 10 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PR/BE/23/228
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — perampanel; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perampanel Tablets (Experimental): Perampanel 10mg Tablets
  Interventions: Drug: Perampanel 10 MG
- Fycompa film-coated tablets (Active Comparator): Fycompa 10mg film-coated tablets (Perampanel 10mg)
  Interventions: Drug: Fycompa 10Mg Tablet

INTERVENTIONS:
Drug: Perampanel 10 MG — 1 tablet of Perampanel Tablets 10mg
  Arms: Perampanel Tablets
Drug: Fycompa 10Mg Tablet — 1 tablet of Perampanel Tablets 10mg
  Arms: Fycompa film-coated tablets

SUMMARY:
An open-label, balanced, randomized, two treatment, two sequence, two period, two way cross-over, single dose bioequivalence study of Perampanel Tablets 10 mg of Humanis Sağlık A.ġ., Turkey and Fycompa 10 mg film-coated tablets of Eisai GmbH Edmund-Rumpler-Straße 3 60549 Frankfurt am Main Deutschland in normal, healthy, adult, human subjects under fasting condition.

ELIGIBILITY:
Inclusion Criteria:

* Subjects fulfilling the following criteria were included in the study:
* Willing to provide written informed consent for participation in the study, and an ability to comprehend the nature and purpose of the study;
* Willing to be available for the entire study period and to comply protocol requirements;
* Normal, healthy, adult, human subject of 18-45 years (both inclusive) of age;
* Body mass index in the range of 18.50 - 30.00 kg/m2 (both inclusive);
* Normal health status as determined by baseline medical and medication history, at the time of screening and vital signs measurements and physical examination at the time of screening as well as check-in of each study period;
* Normal or clinically non-significant laboratory values as determined by hematological, biochemistry tests and urine analysis;
* Normal or clinically non-significant 12-lead ECG recording;
* Non-smokers and willing to abstain from chewing any tobacco containing products at least 72.00 hours prior to check-in until last sample collection in each study period;
* Non Alcoholic;
* Willing to abstain from xanthine or its derivative containing food or beverages (e.g. chocolates, tea, coffee or cola drinks), at least 48.00 hours prior to check-in until last sample collection in each study period;
* Willing to abstain from grapefruit or its juice at least 72.00 hours prior to check-in until last sample collection in each study period;
* For female subjects:
* Negative urine pregnancy test during screening and negative serum β-hCG test at the time of check-in of each study period;
* Female subjects with child bearing potential or those within their first two years of onset of menopausal syndrome willing to either abstain from sexual intercourse, or should use of acceptable birth control methods for at least 15 days before 1st check-in till 15 days post lastdose / entire study period. [Acceptable birth control methods include barrier methods such as diaphragm/condom with or without spermicide or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy has been performed)].

Exclusion Criteria:

* Subjects with the following criteria were excluded from the study:
* Any medical or surgical conditions, which might significantly interfere with the functioning of gastrointestinal tract and of blood forming organs;
* Significant history or current evidence of malignancy or chronic - infectious, cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic (endocrine), hematological, gastrointestinal, dermatological, immunological or psychiatric diseases, or organ dysfunction;
* Any major illness or hospitalized within 90 days prior to the first check-in;
* Requiring medication for any ailment having enzyme-modifying activity within one month prior to first check-in and throughout the study;
* Use of any depot injection or an implant of any drug within 3 months prior to first check-in and throughout the study;
* History or presence of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
* History of Severe cutaneous adverse reactions (SCARs) including drug reaction with eosinophilia and systemic symptoms(DRESS) and Stevens - Johnson Syndrome (SJS).
* Use of any prescribed medication (including herbal medicines and vitamin supplements) or OTC products within 30 days prior to first check-in and throughout the study;
* History or presence of significant gastric and/or duodenal ulceration;
* Difficulty in swallowing tablets or capsules;
* Use of any recreational drug or history of drug addiction;
* Participated in any clinical investigation requiring repeated blood sampling or have donated blood in past 90 days prior to first check-in;
* Positive urine alcohol and urine drug of abuse tests during check-in of each study period;
* Reactive test for Human Immunodeficiency Virus (HIV) type I/II antibodies or Hepatitis B surface antigen (HBsAg) or Hepatitis C virus antibodies;
* Lactating or nursing female subjects;
* Female subjects using hormonal contraceptive (either oral/implants);
* History of allergy or hypersensitivity intolerance to perampanel or its formulation excipients which, in the opinion of a clinical investigator, would compromise the safety of the subject or the study;
* History of difficulty in accessibility of veins in arms.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2023-11-26 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Maximum concentration obtained (Cmax) | 23 hours
  two-sided 90% CI for the test to reference ratio of the population means is within 80.00% to 125.00% for each of the Ln-transformed data Cmax
AUC from time 0 to last collection time 72 (AUC0-72) | 23 hours
  two-sided 90% CI for the test to reference ratio of the population means is within 80.00% to 125.00% for each of the Ln-transformed data AUC0-72

SECONDARY OUTCOMES:
Time of the maximum measured plasma concentration (Tmax) | 23 hours
  Description Statistics

CONTACTS AND LOCATIONS:
Locations (1):
- Raptim Research Pvt. Ltd.,, Navi Mumbai, India

IPD SHARING:
Plan to Share IPD: No